CLINICAL TRIAL: NCT02897115
Title: STRIKE - Treating Patients With Early Axial Spondyloarthritis to Target - a 1 Year Randomized Controlled Study Taking an Intense Treatment Approach Versus Routine Treatment
Brief Title: A Study Treating Participants With Early Axial Spondyloarthritis (axSpA) Taking an Intense Treatment Approach Versus Routine Treatment
Acronym: STRIKE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to slow recruitment.
Sponsor: AbbVie (Industry)
Collaborators: IST GmbH, Germany (Industry); Hannover Medical School (Other); Improvement by Movement GmbH, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W15-679; 2015-005398-18 (EudraCT Number)
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2018-11

CONDITIONS: Axial Spondyloarthritis
Keywords: Axial Spondyloarthritis; Humira
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Adalimumab; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treat-to-Target (T2T) (Experimental): Participants initially received treatment with any non-steroidal anti-inflammatory drug (NSAID) at full anti-inflammatory dose for 4 weeks. After 4 weeks, if the Ankylosing Spondylitis Disease Activity Score (ASDAS) was ≥ 2.1 or treatment with NSAID 1 was not tolerated, treatment was changed to a second NSAID at full anti-inflammatory dose for 4 weeks. If ASDAS was ≥ 2.1 after 4 weeks of NSAID 2 or treatment with the chosen NSAID was not tolerated, , participants were switched to receive a combination of NSAID and adalimumab 40 mg every other week for up to 48 weeks.
  Interventions: Biological: Adalimumab
- Standard of Care (SOC) (Active Comparator): Participants received treatment as prescribed by their physician according to the local standard of care.
  Interventions: Other: Non-steroidal Anti-inflammatory Drugs (NSAIDs)

INTERVENTIONS:
Biological: Adalimumab — Administered every other week by subcutaneous injection for up to 48 weeks, depending on participants' disease activity.
  Other Names: Humira; ABT-D2E7
  Arms: Treat-to-Target (T2T)
Other: Non-steroidal Anti-inflammatory Drugs (NSAIDs) — ASAS recommended NSAID doses to treat axial spondyloarthritis.
  Other Names: Routine practice
  Arms: Standard of Care (SOC)

SUMMARY:
A study comparing a treat-to-target (T2T) intense treatment approach with routine treatment (Standard of Care [SOC]) in reducing disease activity in participants with axial spondyloarthritis (axSpA).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before start of study-related assessments or procedures
* Diagnosis of axSpA (either ankylosing spondylitis or non-radiographic axSpA) and fulfilling the Assessment of Spondyloarthritis International Society (ASAS) classification criteria for axSpA
* Participants aged ≥ 18 years
* Disease duration < 5 years
* Participants must have a Baseline disease activity as defined by an ASDAS ≥ 2.1 or a Bath AS Disease Activity Index (BASDAI) ≥ 4
* NSAID-naive or not treated with the maximal recommended NSAID dose during the last 2 weeks prior to the Baseline visit
* Participants must never have failed a NSAID taken at maximal recommended dose for 2 weeks or more.

Exclusion Criteria:

* Contraindications for NSAIDs or tumor necrosis factor (TNF) blocker according to local labeling
* If entering the study on concomitant NSAIDs, participants taking the maximal recommended dose during the last 2 weeks prior to the Baseline Visit or have failed or developed intolerance to a NSAID taken at maximal recommended dose for 2 weeks or more at any time
* Prior exposure to any anti-TNF therapy; any biologic therapy with a potential therapeutic impact on SpA, or participant has been treated with any investigational drug of chemical or biologic nature within a minimum of 30 days or five half-lives (whichever is longer) of the drug prior to the Baseline visit.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study planned to enroll approximately 240 participants at 30 sites in Germany. Due to slow enrollment the study was terminated prematurely; at the time the decision to close the study was made 22 subjects were enrolled at 9 sites in Germany.
Groups:
- Treat-to-Target (T2T): Participants initially received treatment with any non-steroidal anti-inflammatory drug (NSAID) at full anti-inflammatory dose for 4 weeks. After 4 weeks, if the Ankylosing Spondylitis Disease Activity Score (ASDAS) was ≥ 2.1 or treatment with NSAID 1 was not tolerated, treatment was changed to a second NSAID at full anti-inflammatory dose for 4 weeks. If ASDAS was ≥ 2.1 after 4 weeks of NSAID 2, participants were switched to receive a combination of NSAID and adalimumab 40 mg every other week for up to 48 weeks.
Period: Overall Study
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Started | 14 | 8
Completed | 3 | 0
Not Completed | 11 | 8
Not completed — Early termination of study by sponsor | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC) | Total
Number analyzed (Participants) | 14 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (9.49) | 29.6 (7.96) | 34.3 (9.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Ankylosing Spondylitis Disease Activity Score (ASDAS) of Inactive Disease at Week 32
Description: ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (C-reactive protein [CRP] or erythrocyte sedimentation rate [ESR]) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and > 3.5 for "very high disease activity." The percentage of participants with ASDAS inactive disease (defined as ASDAS < 1.3) calculated using CRP is reported.
Time Frame: Week 32
Population: Participants with available data at week 32
Measure: Number; unit: percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 5 | 1
percentage of participants | 80.0 | 0.0

2. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions (EQ-5D) Questionnaire
Description: The EQ-5D-3L is a health state utility instrument that evaluates preference for health status (utility). The 5 items in the EQ-5D-3L comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on 3 levels of severity (1: indicating no problem, 2: indicating some/moderate problems, 3: indicating extreme problems). A single preference-weighted health utility index score was calculated by applying country-specific weights, with scores ranging from approximately 0 (death) to 1 (full health).
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 7
units on a scale
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | 0.446 (0.181) | -0.287 (NA) — Cannot be calculated when N=1
  Week 52: number analyzed (Participants) | 1 | 0
  Week 52 | 0.255 (NA) — Cannot be calculated when N=1 |

3. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment - Axial Spondyloarthritis (WPAI-axSpA): Presenteeism
Description: The Work Productivity and Activity Impairment (WPAI) axSpA is an axSpA specific questionnaire consisting of 6 questions, based on patient recall of the previous 7 days. WPAI assesses work time missed due to illness (absenteeism), impairment at work due to health (presenteeism), overall work impairment due to health (an aggregate measure of both absenteeism and presenteeism), and total non-occupational activity impairment due to health. WPAI scores are expressed as impairment percentages, with higher scores indicating worse outcomes. A negative change from baseline indicates improvement.
Time Frame: Baseline, week 32, and week 52
Population: Participants who were employed and with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 11 | 5
percent impairment
  Week 32: number analyzed (Participants) | 3 | 1
  Week 32 | -23.3 (55.1) | 20.0 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment - Axial Spondyloarthritis (WPAI-axSpA): Absenteeism
Description: as for outcome 3
Time Frame: Baseline, week 32, and week 52
Population: Participants who were employed and with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 11 | 6
percent impairment
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | -100.0 (NA) — Could not be calculated when N=1 | 25.0 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 1 | 0
  Week 52 | -100.0 (NA) — Could not be calculated when N=1 |

5. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment - Axial Spondyloarthritis (WPAI-axSpA): Total Work Productivity Impairment
Description: as for outcome 3
Time Frame: Baseline, week 32, and week 52
Population: Participants who were employed and with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 11 | 5
percent impairment
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | -90.0 (NA) — Could not be calculated when N=1 | 27.5 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 1 | 0
  Week 52 | -80.0 (NA) — Could not be calculated when N=1 |

6. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment - Axial Spondyloarthritis (WPAI-axSpA): Total Activity Impairment
Description: as for outcome 3
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 6
percent impairment
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | -36.0 (15.2) | 30.0 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 1 | 0
  Week 52 | -30.0 (NA) — Could not be calculated when N=1 |

7. Secondary Outcome: Change From Baseline in Assessment of Spondyloarthritis International Society (ASAS) Health Index (HI)
Description: The ASAS HI measures functioning and health across 17 aspects of health in patients with AS, including pain, emotional functions, sleep, sexual function, mobility, self care, and community life. The ASAS HI consists of 17 questions, each answered by the participant as agree (1) or disagree (0). The responses to the 17 dichotomous items are summed up to give a total score ranging from 0 to 17, with a lower score indicating a better and a higher score indicating an inferior health status.
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 13 | 7
score on a scale
  Week 32: number analyzed (Participants) | 4 | 1
  Week 32 | -4.00 (2.45) | 3.00 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 1 | 0
  Week 52 | -3.00 (NA) — Could not be calculated when N=1 |

8. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Disease Activity Index
Description: The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) assesses disease activity by asking the participant to answer 6 questions (each on a 10 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For 5 questions (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10 where lower scores indicate less disease activity.
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
score on a scale
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | -3.96 (1.68) | 3.20 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | -1.83 (3.18) |

9. Secondary Outcome: Percentage of Participants Achieving a BASDAI 50 Response
Description: The BASDAI assesses disease activity by asking the participant to answer 6 questions (each on a 10 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For 5 questions (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10. Lower scores indicate less disease activity.
  A BASDAI 50 response is defined as improvement of 50% or more from baseline in BASDAI score.
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Number; unit: percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
percentage of participants
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | 60.0 | 0.0
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | 33.3 |

10. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: The Bath Ankylosing Spondylitis Functional Index (BASFI) is a validated index to determine the degree of functional limitation in patients with AS. BASFI consists of 10 questions assessing participants' ability to perform activities, on a numeric rating scale (NRS) ranging from 0 (easy to perform an activity) to 10 (impossible to perform an activity). The overall score is the mean of the 10 items and ranges from 0 (best) to 10 (worst).
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
score on a scale
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | -2.46 (2.14) | -1.50 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -1.40 (0.849) |

11. Secondary Outcome: Change From Baseline in ASDAS(CRP)
Description: ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP or ESR) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and > 3.5 for "very high disease activity." Change from baseline in ASDAS calculated using CRP is reported.
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 7
score on a scale
  Week 32: number analyzed (Participants) | 5 | 0
  Week 32 | -1.29 (0.833) |
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | -0.654 (1.22) |

12. Secondary Outcome: Percentage of Participants Achieving ASDAS(CRP) Major Improvement
Description: ASDAS Major Improvement is defined as a change from baseline ≤ -2.0. ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP or ESR) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and > 3.5 for "very high disease activity." The percentage of participants with major improvement in ASDAS calculated using CRP is reported.
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Number; unit: percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 7
percentage of participants
  Week 32: number analyzed (Participants) | 5 | 0
  Week 32 | 20.0 |
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | 33.3 |

13. Secondary Outcome: Percentage of Participants Achieving ASDAS(CRP) Clinically Important Improvement
Description: ASDAS clinically important improvement is defined as a change from baseline ≤ -1.1.
  ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP or ESR) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and > 3.5 for "very high disease activity." The percentage of participants with clinically important improvement in ASDAS calculated using CRP is reported.
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Number; unit: percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 7
percentage of participants
  Week 32: number analyzed (Participants) | 5 | 0
  Week 32 | 60.0 |
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | 33.3 |

14. Secondary Outcome: Percentage of Participants With ASDAS Inactive Disease at Week 52
Description: ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP or ESR) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and > 3.5 for "very high disease activity." The percentage of participants with ASDAS inactive disease (defined as ASDAS < 1.3) calculated using CRP is reported.
Time Frame: Week 52
Population: Participants with available data at week 52
Measure: Number; unit: percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 3 | 0
percentage of participants | 33.3 |

15. Secondary Outcome: Percentage of Participants With ASDAS Low Disease Activity
Description: ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP or ESR) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and > 3.5 for "very high disease activity." The percentage of participants with ASDAS low disease activity (defined as ASDAS < 2.1) calculated using CRP is reported.
Time Frame: Week 32 and week 52
Population: Participants with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 7
percentage of participants
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | 80.0 | 0.0
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | 66.7 |

16. Secondary Outcome: Percentage of Participants With ASDAS Moderate Disease Activity
Description: ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP or ESR) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and > 3.5 for "very high disease activity." The percentage of participants with ASDAS moderate disease activity (defined as an ASDAS ≥ 1.3 to < 2.1) calculated using CRP is reported.
Time Frame: Week 32 and week 52
Population: Participants with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 7
percentage of participants
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | 0.0 | 0.0
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | 33.3 |

17. Secondary Outcome: Percentage of Participants With ASDAS High Disease Activity
Description: ASDAS high disease activity is defined as an ASDAS ≥ 2.1 to < 3.5. ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP or ESR) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and > 3.5 for "very high disease activity." The percentage of participants with high disease activity (defined as an ASDAS ≥ 2.1 to < 3.5) calculated using CRP is reported.
Time Frame: Week 32 and week 52
Population: Participants with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 7
percentage of participants
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | 20.0 | 100.0
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | 33.3 |

18. Secondary Outcome: Percentage of Participants With ASDAS Very High Disease Activity
Description: ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP or ESR) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and > 3.5 for "very high disease activity." The percentage of participants with very high disease activity (defined as an ASDAS > 3.5) calculated using CRP is reported
Time Frame: Week 32 and week 52
Population: Participants with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 7
percentage of participants
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | 0.0 | 0.0
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | 0.0 |

19. Secondary Outcome: Percentage of Participants Achieving an Assessment of Spondyloarthritis International Society (ASAS) 20 Response
Description: ASAS20 response was defined as improvement of ≥ 20% relative to baseline and absolute improvement of ≥ 1 unit (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration (defined as a worsening of ≥ 20% and a net worsening of ≥ 1 unit) in the potential remaining domain:
  * Patient's Global Assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (none) to 10 (severe);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Number; unit: percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 7
percentage of participants
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | 40.0 | 0.0
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | 50.0 |

20. Secondary Outcome: Percentage of Participants Achieving an ASAS 40 Response
Description: ASAS40 response was defined as improvement of ≥ 40% relative to baseline and absolute improvement of ≥ 2 units (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration in the potential remaining domain:
  * Patient's Global Assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (none) to 10 (severe);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Number; unit: percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 7
percentage of participants
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | 20.0 | 0.0
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | 50.0 |

21. Secondary Outcome: Percentage of Participants Achieving ASAS Partial Remission
Description: ASAS partial remission is defined as an absolute score of ≤ 2 units on a 0 to 10 scale for each of the four following domains:
  * Patient's Global Assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (none) to 10 (severe);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Week 32 and week 52
Population: Participants with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 7
percentage of participants
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | 0.0 | 0.0
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | 50.0 |

22. Secondary Outcome: Change From Baseline in Active Inflammation of the Sacroiliac Joints and Spine
Description: Active inflammation of the sacroiliac (SI) joints as well as the cervical, thoracic and lumbar regions of the spine was assessed using magnetic resonance imaging (MRI). Images were scored by a central reader according to the Berlin MRI Score on a grading scale from 0 to 3, where Grade 0 indicates no active inflammation and Grade 3 indicates > 66% inflammation of the sacroiliac joints or > 50% active inflammation in the spine.
Time Frame: Baseline and week 52
Population: The study terminated early due to slow enrollment and no data were collected.
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity
Description: The Physician's Global Assessment of Disease Activity was assessed using an NRS from 0 (no disease activity) to 10 (severe disease activity).
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
score on a scale
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | -4.00 (1.41) | 1.00 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | -2.00 (3.00) |

24. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity
Description: The Patient's Global Assessment of Disease Activity was assessed using an NRS from 0 (no disease activity) to 10 (very severe disease activity).
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
score on a scale
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | -2.20 (3.90) | 4.00 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | -1.00 (3.61) |

25. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Pain
Description: The Patient's Global Assessment of Pain was assessed on a NRS from 0 (no pain) to 10 (pain as bad as it could be).
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
score on a scale
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | -1.60 (4.28) | 3.00 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | -0.333 (2.08) |

26. Secondary Outcome: Change From Baseline in Swollen Joint Count
Description: An assessment of 66 joints was performed by physical examination of each joint. The swollen joint count is the number of joints assessed as swollen (0 to 66).
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
swollen joints
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | 0.0000 (0.0000) | 0.0000 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | 0.333 (0.577) |

27. Secondary Outcome: Change From Baseline in Tender Joint Count
Description: An assessment of 68 joints was performed by physical examination of each joint. The tender joint count is the number of joints assessed as tender (0 to 68).
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
tender joints
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | -3.40 (5.98) | 1.00 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | -6.33 (6.66) |

28. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES)
Description: The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at 13 entheses (sites where tendons or ligaments insert into the bone). All sites were scored as 0 (absent) or 1 (present). The MASES is the sum of all site scores (from 0 to 13).
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
score on a scale
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | -0.800 (1.79) | 0.0000 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | 0.333 (1.53) |

29. Secondary Outcome: Change From Baseline in Dactylitis Count
Description: Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as 0 for no dactylitis or 1 for dactylitis present. The dactylitis count, ranging from 0 to 20, is the total number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: digits with dactylitis
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
digits with dactylitis
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | 0.0000 (0.0000) | 0.0000 (NA) — Could not be calculated when N=0
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | 0.0000 (0.0000) |

30. Secondary Outcome: Change From Baseline in the Erythrocyte Sedimentation Rate (ESR)
Description: Erythrocyte sedimentation rate measures the rate of fall (sedimentation) of erythrocytes (red blood cells) in a sample of blood that has been placed into a tall, thin, vertical tube as an indirect measure of the degree of inflammation present in the body.
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
mm/hour
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | -2.60 (3.05) | 0.0000 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | -4.00 (3.46) |

31. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP)
Description: CRP is an acute phase reactant is a blood test marker for inflammation in the body. CRP levels rise in response to inflammation.
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
mg/L
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | -4.47 (4.38) | -1.00 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | -3.47 (6.00) |

32. Secondary Outcome: Change From Baseline in Linear Bath Ankylosing Spondylitis Metrology Index (BASMIlin)
Description: The linear Bath Ankylosing Spondylitis Metrology Index (BASMIlin) is a composite score based on 5 direct measurements of spinal mobility: lateral lumbar flexion, tragus-to-wall distance, lumbar flexion, intermalleolar distance, and cervical rotation angle. The total score ranges from 0 to 10, where higher scores indicate more limited mobility.
Time Frame: Baseline, week 32, and week 52
Population: Participants with available data at baseline and each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
score on a scale
  Week 32: number analyzed (Participants) | 5 | 1
  Week 32 | -1.00 (0.632) | -1.10 (NA) — Could not be calculated when N=1
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -1.20 (0.944) |

33. Secondary Outcome: Number of Participants With New Onset Anterior Uveitis
Description: Anterior uveitis is an inflammation of the middle layer of the eye. which includes the iris (colored part of the eye) and the adjacent tissue, known as the ciliary body.
Time Frame: Up to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treat-to-Target (T2T) | Standard of Care (SOC)
Number analyzed (Participants) | 14 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Arm/Group | Standard of Care (SOC) | Treat-to-Target (T2T)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/14
Other Adverse Events (participants affected / at risk) | 6/8 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (SOC) (N=8) | Treat-to-Target (T2T) (N=14)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=8) | Treat-to-Target (T2T) (N=14)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 3 (4)
ANAL FISSURE (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (2)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 2 (2)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (2)
CYSTITIS (Infections and infestations) | 1 (1) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 4 (4)
PULPITIS DENTAL (Infections and infestations) | 0 (0) | 1 (1)
RHINITIS (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST-TRAUMATIC NECK SYNDROME (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
AXIAL SPONDYLOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
DYSAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (2)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (2)
MOOD ALTERED (Psychiatric disorders) | 1 (1) | 0 (0)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VULVOVAGINAL INFLAMMATION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT02897115/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT02897115/SAP_001.pdf